CLINICAL TRIAL: NCT00004401
Title: Study of Human Botulism Immunoglobulin in Infants With Botulism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: California Department of Health Services (Other)
Organization: FDA Office of Orphan Products Development (U.S. Federal Agency)
Masking: None | Purpose: Treatment
Other Study IDs: 199/13253; CDHS-FDU000476
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2000-03

CONDITIONS: Infant Botulism; Botulism
Keywords: bacterial infection; clostridium infection; immunologic disorders and infectious disorders; infant botulism; rare disease
MeSH Terms: conditions — Botulism; Bacterial Infections; Clostridium Infections; Immune System Diseases; Communicable Diseases; Rare Diseases | interventions — botulism immune globulin

INTERVENTIONS:
Drug: botulism immune globulin

SUMMARY:
OBJECTIVES: I. Determine the safety of human botulism immune globulin (BIG) in patients with infant botulism by monitoring side effects (e.g., rash, fever, hypotension, and anaphylaxis).

II. Assess the efficacy of BIG in these patients by monitoring disease severity, incidence of complications (respiratory arrest, aspiration, pneumonia, etc.), and length of hospital stay.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is an open label, multicenter study. Patients should begin therapy within 72 hours of hospital admission, but may receive human botulism immunoglobulin (BIG) in certain circumstances after 72 hours. Patients receive (BIG) IV. Patients are monitored for side effects, disease severity, complications, and length of hospital stay.

Patients are followed at 2 weeks after treatment, then every 4 weeks for 6 months.

Completion date provided represents the completion date of the grant per OOPD records

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

* Clinical diagnosis of infant botulism in previously healthy infant
* Bulbar palsies
* Constipated Lethargy
* Diminished head control
* Poor feeding
* Generalized weakness and hypotonia
* Weak cry
* Afebrile (unless secondary infection present)
* Subacute to acute onset
* Normal electrolytes
* Any patient eligible provided no treatment available for life-threatening condition

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 1998-01; Study Completion 1998-06

CONTACTS AND LOCATIONS:
Overall Officials: Stephen S. Arnon, Study Chair — California Department of Health Services
Locations (1):
- California Department of Health Services, Berkeley, California, United States